CLINICAL TRIAL: NCT02721758
Title: Design and Evaluation of a Brief Motivational Intervention to Promote Enrolment in Outpatient Cardiac Rehabilitation
Brief Title: Understanding and Promoting Health Behaviour Change Amid Transition to Cardiac Rehabilitation
Acronym: UPBeAT-CR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Tavis S. Campbell, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REB14-1213
Record Dates: First submitted 2016-03-18; First posted 2016-03-29 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Patient Compliance
Keywords: Motivational Interviewing; Health Behavior; Cardiac Rehabilitation
MeSH Terms: conditions — Patient Compliance; Health Behavior

ARMS (2):
- Brief Motivational Intervention (Experimental): Single, 60-minute, manualized behavioural intervention designed to support cardiac rehabilitation enrollment, informed by principles of motivational interviewing
  Interventions: Behavioral: Brief Motivational Intervention
- Usual Care (No Intervention): Standard encouragement to enroll in cardiac rehabilitation, and meeting with a researcher to complete study questionnaires

INTERVENTIONS:
Behavioral: Brief Motivational Intervention
  Arms: Brief Motivational Intervention

SUMMARY:
The purpose of this study was to test whether a brief motivational intervention is associated with enrollment in cardiac rehabilitation.

DETAILED DESCRIPTION:
Cardiac rehabilitation programs help reduce morbidity and mortality following a cardiac event, but only a subset of referred patients chooses to participate. An intervention based on principles of motivational interviewing may help resolve individuals' ambivalence about cardiac rehabilitation. The primary aim is to evaluate the efficacy of a brief motivational intervention (MI) for enhancing intention to enroll in cardiac rehabilitation compared to a usual care (UC) control condition among patients referred to cardiac rehabilitation. It is hypothesized that patients in the MI condition will report greater intention to enroll in cardiac rehabilitation compared to patients in UC. A small-scale feasibility trial will include patients (n = 100) with acute coronary syndrome who are referred to a standard 12-week exercise-based cardiac rehabilitation program in Calgary, Canada. Patients will be randomly assigned to MI or UC. The primary outcome will be self-reported intention to attend cardiac rehabilitation. Secondary outcomes will include beliefs about cardiac rehabilitation, exercise self-efficacy, perceived barriers, and cardiac rehabilitation enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Referred to and eligible for outpatient, exercise-based cardiac rehabilitation; confirmed acute coronary syndrome; English-speaking; able to complete study prior to first scheduled cardiac rehabilitation appointment

Exclusion Criteria:

* Cognitive or hearing impairment that would interfere with study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Intention to Attend Cardiac Rehabilitation Scale (adapted from Blanchard et al., 2002) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  Intention to attend cardiac rehabilitation will be assessed using the average of two self-report items: (1) "My goal is to attend ___ exercise classes at cardiac rehabilitation" with responses ranging from 1 (no exercise classes) to 7 (some exercise classes) and (2) "I intend to attend scheduled classes during cardiac rehabilitation" with responses ranging from 1 (strongly disagree) to 7 (strongly agree).
  Blanchard, C. M., Courneya, K. S., Rodgers, W. M., Daub, B., & Knapik, G. (2002). Determinants of exercise intention and behavior during and after phase 2 cardiac rehabilitation: An application of the theory of planned behavior. Rehabilitation Psychology, 47(3), 308-323.

SECONDARY OUTCOMES:
Cardiac Rehabilitation Enrollment (attendance at ≥1 appointment; chart review) | 60 days after initial referral to cardiac rehabilitation program
  Participation in cardiac rehabilitation will be confirmed by chart review 60 days after referral. Non-enrollment will be defined as (a) explicitly declining interest in CR participation, (b) not attending the initial scheduled exercise appointment within 60 days of referral, or (c) inability to be contacted by program staff within 60 days of referral to cardiac rehabilitation.
Beliefs About Cardiac Rehabilitation Scale (BACR; Cooper et al., 2007) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  The BACR is a 13-item questionnaire that evaluates patients' beliefs regarding CR. Items are rated on a 5-point Likert-type scale, ranging from "strongly disagree" to "strongly agree." Items are summed to provide a score on each of four subscales: perceived necessity, concerns about exercise, practical barriers, and perceived suitability.
  Cooper, A. F., Weinman, J., Hankins, M., Jackson, G., & Horne, R. (2007). Assessing patients' beliefs about cardiac rehabilitation as a basis for predicting attendance after acute myocardial infarction. Heart (British Cardiac Society), 93(1), 53-8. doi:10.1136/hrt.2005.081299
Multidimensional Self-Efficacy for Exercise Scale (Rodgers et al., 2008) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  The MSES is a 9-item questionnaire that evaluates exercise self-efficacy in three domains: task (e.g., ability to follow directions to complete exercise), coping (e.g., ability to exercise when feeling discomfort from exercise), and scheduling (e.g. ability to fit exercise into daily routine). Items are rated from 0 (not at all confident) to 100 (completely confident), and averaged in each domain.
  Rodgers, W. M., Wilson, P. M., Hall, C. R., Fraser, S. N., & Murray, T. C. (2008). Evidence for a multidimensional self-efficacy for exercise scale. Research Quarterly for Exercise and Sport, 79(2), 222-34.
Cardiac Rehabilitation Barriers Scale (CRBS; Shanmugasegaram et al., 2012) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  The CRBS is a 21-item questionnaire designed to assess perceptions of patient, provider, and health system barriers to CR participation. Items are rated on 5-point Likert-type scales ranging from "strongly disagree" to "strongly agree," and are averaged to provide a total score, with higher scores indicating greater perceived barriers. Totals are also calculated for four subscales: perceived need/healthcare factors, logistical factors, work/time conflicts, and comorbidities/functional status.
  Shanmugasegaram, S., Gagliese, L., Oh, P., Stewart, D. E., Brister, S. J., Chan, V., & Grace, S. L. (2012). Psychometric validation of the Cardiac Rehabilitation Barriers Scale. Clinical Rehabilitation, 26(2), 152-64. doi:10.1177/0269215511410579

OTHER OUTCOMES:
ENRICHD Social Support Instrument (ESSI; Mitchell et al., 2003) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  The ESSI is a 7-item questionnaire designed to assess social support in patients post-myocardial infarction. Items are rated from 1 (none of the time) to 5 (all of the time), and are summed to provide a total score, with higher scores indicating more social support.
  Mitchell, P. H., Powell, L., Blumenthal, J., Norten, J., Ironson, G., Pitula, C. R., ... & Berkman, L. F. (2003). A short social support measure for patients recovering from myocardial infarction: the ENRICHD Social Support Inventory. Journal of Cardiopulmonary Rehabilitation and Prevention, 23(6), 398-403.
Brief Illness Perceptions Questionnaire (BIPQ; Broadbent et al., 2006) | At least 1 day after receiving MI or UC but prior to enrollment in cardiac rehabilitation (average 7 days)
  The BIPQ is an 8-item questionnaire that assesses cognitive and emotional representations of illness. It evaluates perceived consequences, timelines, personal/treatment control, symptoms, concern, understanding, and emotional consequences associated with the illness. Items are summed to provide a total score, with higher scores indicating greater perceived threat of the illness.
  Broadbent, E., Petrie, K. J., Main, J., & Weinman, J. (2006). The brief illness perception questionnaire. Journal of Psychosomatic Research, 60(6), 631-7. doi:10.1016/j.jpsychores.2005.10.020
Cardiac rehabilitation adherence (# of cardiac rehabilitation sessions attended; chart review) | Following a 12-week cardiac rehabilitation program
  Number of cardiac rehabilitation sessions attended (out of a total possible 24 scheduled sessions)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, University of Calgary, Calgary, Alberta, Canada